CLINICAL TRIAL: NCT00633009
Title: A Blinded, Placebo Controlled Study Evaluating Safety, False-Positive Reactions and Sensitizing Properties of Leishmania Tropica Skin Test Antigen (LtSTA)
Brief Title: Safety, False-Positive Reactions and Sensitizing Properties of Leishmania Tropica Skin Test Antigen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nielsen BioSciences, Inc. (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: LtSTA-08
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Results first posted 2012-12-06 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-10

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Leishmaniasis; Delayed-Type Hypersensitivity (DTH); Skin Test; Conversion; Prior exposure to Leishmania major
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis; Hypersensitivity, Delayed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LtSTA 15 ug (Active Comparator): Naive volunteers tested with 15 ug injection of LtSTA. Participants were skin tested on visits 3, 6 and 9 of the study. The results of the skin tests were read after 48 hours (+/- 6 hours) on visits 4, 7 and 10. A final evaluation was performed on visit 11, fourteen days after visit 10.
  Interventions: Biological: Leishmania tropica Skin Test Antigen (LtSTA); Biological: Leishmania tropica Skin Test Antigen Placebo (Placebo)
- LtSTA 30 ug (Active Comparator): Naive volunteers tested with 30 ug injection of LtSTA.Participants were skin tested on visits 3, 6 and 9 of the study. The results of the skin testes were read after 48 hours (+/- 6 hours) on visits 4, 7 and 10. A final evaluation was performed on visit 11, fourteen days after visit 10.
  Interventions: Biological: Leishmania tropica Skin Test Antigen (LtSTA); Biological: Leishmania tropica Skin Test Antigen Placebo (Placebo)
- LtSTA 50 ug (Active Comparator): Naive volunteers tested with 50 ug injection of LtSTA.Participants were skin tested on visits 3, 6 and 9 of the study. The results of the skin testes were read after 48 hours (+/- 6 hours) on visits 4, 7 and 10. A final evaluation was performed on visit 11, fourteen days after visit 10.
  Interventions: Biological: Leishmania tropica Skin Test Antigen (LtSTA); Biological: Leishmania tropica Skin Test Antigen Placebo (Placebo)

INTERVENTIONS:
Biological: Leishmania tropica Skin Test Antigen (LtSTA) — Administer 15 ug, 30 ug or 50 ug of LtSTA into DTH positive volunteers. Repeat drug administration 30 days after initial injection and 60 days after initial injection. Read and interpret reaction 48 hours after each injection. Observe subjects for conversion or adverse reaction.
Biological: Leishmania tropica Skin Test Antigen Placebo (Placebo) — Administer Placebo concurrently with 15 ug, 30 ug and 50 ug doses of LtSTA. Read and interpret the reaction 48 hours after injection. Observe subjects for reaction to Placebo

SUMMARY:
The efficacy of LtSTA as a skin test antigen depends upon the sensitivity and specificity of the product. This study has been designed to measure the skin test responses to 15, 30, or 50µg doses of LtSTA. The measurements of non-specific reactivity due to components of the antigen solution and the product's ability to sensitize lymphocytes of Leishmania naïve persons when administered intradermally. The presence or absence of a local inflammatory response to the first skin test with each of three doses of LtSTA will provide insight on the specificity of the antigen in a naïve population. The local inflammatory response to LtSTA following the first and second repeat skin tests will indicate if the antigen is sensitizing after intradermal administration.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female in good health;
* Age 18 - 60 years;
* No past history of leishmaniasis or prior participation in a Leishmania study;
* No prior skin test with a Leishmania antigen;
* No occupational, residential, or travel exposure to Leishmania;
* Positive Candin® or Trichophyton skin test (>= 5 mm induration).

Exclusion Criteria:

* History of adult atopic dermatitis, contact dermatitis to multiple agents, unexplained urticaria, or asthma;
* Active allergic rhinitis or conjunctivitis;
* History of allergy or reactions to phenol, polysorbate 80, or glycerol;
* Medications: currently taking (within the last month) antihistamines or recent history of taking (within the last 1 year) corticosteroids, immunosuppressants;
* Splenectomy;
* Active medical disease*;

  *Active Medical Disease: Any active physical or psychiatric condition that may increase the risks associated with participation in the study or interferes with the interpretation of study results. Included chronic medical illnesses are cardiovascular disease, renal insufficiency, chronic respiratory illness, cirrhosis, chronic hepatitis, chronic pancreatitis, chronic diarrhea, malnutrition, malignancy, autoimmune disease, and asthma.
* Pregnancy or lactating;
* Immunization within 4 weeks;
* History of leishmaniasis;
* Occupational exposure to Leishmania;
* Prior participation in a Leishmania study;
* Prior skin test with Leishmania antigen;
* Travel history to Leishmania endemic areas;
* Abnormal screening lab results;
* Keloid scar formation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry S Nielsen, Ph.D., Study Director — Nielsen BioSciences, Inc.; Donald M Brandon, M.D., Principal Investigator — California Research Foundation
Locations (1):
- California Research Foundation, San Diego, California, United States

REFERENCES:
- See also: Allermed Laboratories, Inc. — http://www.allermed.com

RESULTS

PARTICIPANT FLOW:
Groups:
- 15 ug Study Group: Naive volunteers tested with 15 ug injection of LtSTA. Participants were skin tested on visits 3, 6 and 9 of the study. The results of the skin tests were read after 48 hours (+/- 6 hours) on visits 4, 7 and 10. A final evaluation was performed on visit 11, fourteen days after visit 10. All participants received a placebo skin test concurrently with active drug.
- 30 ug Study Group: Naive volunteers tested with 30 ug injection of LtSTA.Participants were skin tested on visits 3, 6 and 9 of the study. The results of the skin tests were read after 48 hours (+/- 6 hours) on visits 4, 7 and 10. A final evaluation was performed on visit 11, fourteen days after visit 10.All participants received a placebo skin test concurrently with active drug.
- 50 ug Study Group: Naive volunteers tested with 50 ug injection of LtSTA.Participants were skin tested on visits 3, 6 and 9 of the study. The results of the skin tests were read after 48 hours (+/- 6 hours) on visits 4, 7 and 10. A final evaluation was performed on visit 11, fourteen days after visit 10.All participants received a placebo skin test concurrently with active drug.
Period: Overall Study
Arm/Group | 15 ug Study Group | 30 ug Study Group | 50 ug Study Group
Started | 12 | 27 | 11
Completed | 8 | 23 | 10
Not Completed | 4 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- 15 ug Study Group: Naive volunteers tested with 15 ug injection of LtSTA. Participants were skin tested on visits 3, 6 and 9 of the study. The results of the skin tests were read after 48 hours (+/- 6 hours) on visits 4, 7 and 10. A final evaluation was performed on visit 11, fourteen days after visit 10.
- 30 ug Study Group: Naive volunteers tested with 30 ug injection of LtSTA.Participants were skin tested on visits 3, 6 and 9 of the study. The results of the skin tests were read after 48 hours (+/- 6 hours) on visits 4, 7 and 10. A final evaluation was performed on visit 11, fourteen days after visit 10.
- 50 ug Study Group: Naive volunteers tested with 50 ug injection of LtSTA.Participants were skin tested on visits 3, 6 and 9 of the study. The results of the skin tests were read after 48 hours (+/- 6 hours) on visits 4, 7 and 10. A final evaluation was performed on visit 11, fourteen days after visit 10.
- Total: Total of all reporting groups
Arm/Group | 15 ug Study Group | 30 ug Study Group | 50 ug Study Group | Total
Number analyzed (Participants) | 12 | 27 | 11 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 3 | 0 | 3
  Between 18 and 65 years | 12 | 24 | 11 | 47
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34 (11) | 28 (12) | 35 (13) | 31 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 4 | 23
  Male | 3 | 17 | 7 | 27
Region of Enrollment [Number; unit: participants]
  United States | 12 | 27 | 11 | 50

OUTCOME MEASURES:

1. Primary Outcome: Sensitizing Effects of LtSTA in Leishmania Naive Adults
Description: Skin test response of subjects in the trial were evaluated 48 hours post injection after each of three skin test given at 30 day intervals in naive individuals (no exposure to the Leishmania organism). (Actual times 0, 30 and 60 days).The outcome measure was designated as number of participants who became sensitized to the Leishmania antigen. This is defined as those participants that had a negative skin test result, followed by a positive response in a subsequent skin test without having been exposed to the Leishmania organism.
Time Frame: 62 days
Population: Number of participants completed.
Measure: Number; unit: participants
Arm/Group | 15 ug Study Group | 30 ug Study Group | 50 ug Study Group
Number analyzed (Participants) | 8 | 23 | 10
participants | 8 | 22 | 9

2. Secondary Outcome: The Safety of 15, 30 and 50µg/0.1mL Doses of LtSTA in Healthy Adult Volunteers Who Have Had no Known Previous Exposure to Leishmania Parasites
Description: Local and systemic events following skin test. Local: burning, itching, pain. Systemic: Body aches, dizziness, nausea, weakness.
Time Frame: 74 days
Measure: Number; unit: No. of participants with reactions
Arm/Group | 15 ug Study Group | 30 ug Study Group | 50 ug Study Group
Number analyzed (Participants) | 12 | 27 | 11
No. of participants with reactions | 3 | 6 | 2

ADVERSE EVENTS:
Time Frame: 106 Days
Description: Injections of LtSTA were given 3 times over a 90 day period at 30 days +/- 7 days. Final skin test readings were taken at 48 hours after the third injection. Adverse event data were collected for an additional 14 days.
Arm/Group | 15 ug Study Group | 30 ug Study Group | 50 ug Study Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/27 | 0/11
Other Adverse Events (participants affected / at risk) | 3/12 | 6/27 | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 ug Study Group (N=12) | 30 ug Study Group (N=27) | 50 ug Study Group (N=11)
Itching (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 2 (2) — Reported in diary.
Burning (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) — Reported in diary.
Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) — Reported in diary.
Body Aches (General disorders) | 1 (1) | 0 (0) | 1 (1) — Reported in diary.
Weakness (General disorders) | 1 (1) | 0 (0) | 0 (0) — Reported in diary.
Dizziness (General disorders) | 2 (2) | 0 (0) | 0 (0) — Reported in diary.
Nausea (General disorders) | 2 (2) | 0 (0) | 0 (0) — Reported in diary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes